CLINICAL TRIAL: NCT04432883
Title: Targeted Transcranial Direct Current Stimulation to Enhance Speech-Language Treatment Outcome in Persons With Chronic Post-Stroke Aphasia
Brief Title: Targeted TDCS to Enhance Speech-Language Treatment Outcome in Persons With Chronic Post-Stroke Aphasia.
Acronym: AphasiatDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jessica Richardson, Assistant Professor: SOM Neurosurgery, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNM HRRC #16-091; 1P20GM109089-01A1 (NIH); R01DC018282 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2020-06-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Aphasia
Keywords: Stroke; Aphasia; brain stimulation; communication problems; speech and language therapy
MeSH Terms: conditions — Stroke; Aphasia; Communication Disorders | interventions — Language Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental: Active cathodal tDCS + Speech-language training (Active Comparator): In this arm, 31 patients with stroke induced Aphasia will undergo 15 sessions of active tDCS (x 30 minutes of stimulation) combined with 1 hour simultaneous speech-language training on consecutive weekdays.
  Interventions: Device: Active Comparator: Experimental: Active cathodal tDCS + language training
- Comparator: Placebo cathodal tDCS + Speech-language training (Sham Comparator): In this arm, 31 patients with stroke induced Aphasia will undergo 15 sessions of sham tDCS (x 30 minutes sham) combined with 1 hour simultaneous speech-language training on consecutive weekdays..
  Interventions: Behavioral: Sham Comparator: Placebo cathodal tDCS + Speech and language

INTERVENTIONS:
Device: Active Comparator: Experimental: Active cathodal tDCS + language training — Cathodal tDCS raises neuronal membrane potentials, leading to decreased probability of depolarization from incoming stimuli.
  Speech and Language training involves a combined semantic feature analysis and phonological components analysis treatment.
  Other Names: Behavioral: Speech and Language Training
  Arms: Experimental: Active cathodal tDCS + Speech-language training
Behavioral: Sham Comparator: Placebo cathodal tDCS + Speech and language — Speech and Language training involves a combined semantic feature analysis and phonological components analysis treatment. .
  Arms: Comparator: Placebo cathodal tDCS + Speech-language training

SUMMARY:
62 patients who are one year post stroke and have Aphasia as a result of that stroke will be recruited. Participants will have 4 assessment sessions and 15 treatment sessions. The TDCS will be to right Inferior Frontal Gyrus (IFG) (25 active, 25 sham) for 15 days. A combined semantic feature analysis/phonological components analysis treatment will be paired with the stimulation. Two assessment sessions will be pretreatment, 1 session immediately post-treatment, and 1 session at 3 months follow-up.

DETAILED DESCRIPTION:
Our long-term goal is to develop safe and effective treatments for the communication problems of Aphasia due to stroke that restore patients to higher levels of functioning, decrease disability, and promote higher quality of life. While language therapy for aphasia is effective, improvements are typically slow, and gains may be small. Noninvasive brain stimulation has been suggested as a method to enhance outcomes from language therapy. This study will examine whether outcomes for language therapy with brain stimulation are different from outcomes for language therapy without brain stimulation in people with aphasia. Our central hypotheses are (1) targeted right hemisphere HDtDCS (RH-HD-tDCS) administered in combination with language treatment will result in greater changes in naming accuracy than language treatment with the sham RH-HD-tDCS (2) RH-HD-tDCS plus language treatment will result in greater increases in communication within the affected hemisphere compared to language treatment plus sham RH-HD-tDCS (3) RH-HD-tDCS plus language treatment will result in greater increases in perilesional areas working together immediately post-treatment compared to language treatment plus sham RH-HD-tDCS

ELIGIBILITY:
Inclusion Criteria:

1. aged 25-85
2. must be greater than 6 months post-stroke
3. must have a diagnosis of aphasia based on impaired performance on the Western Aphasia Battery-Revised, Boston Naming Test, or during discourse production
4. must be left-hemisphere dominant as demonstrated by aphasia onset subsequent to left hemisphere damage
5. must be stimulable for naming

Exclusion Criteria:

1. comorbid neurological disease.
2. damage to the anterior right hemisphere.
3. significant mood disorder.
4. substance/alcohol dependence or abuse within the past year
5. presence of any implanted electrical device or contraindications to tDCS or MRI
6. recent medical instability (within 4 weeks)
7. pregnancy

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Picture Naming of trained items | 3 months
  Change in naming of pictures of trained items; 60 pictured items; higher score indicates improvement
Naming Response Time of trained items Scales - IV (WAIS-IV; Wechsler, Coalson, & Railford, 2008) | 3 months
  Change in response time of naming of pictures of trained items; 0-20 seconds, decreased response time indicates improvement Scales - IV (WAIS-IV; Wechsler, Coalson, & Railford, 2008)
Naming Efficiency of trained items | 3 months
  Change in efficiency of naming of pictures of trained items; median response time divided by proportion correct naming; smaller numbers indicate greater efficiency

SECONDARY OUTCOMES:
Discourse informativeness - Main Concept Production | 3 months
  Change in discourse informativeness as measured by main concept scores; increased values indicate improvement
Efficiency of discourse informativeness - Main Concept Production | 3 months
  Change in efficiency of discourse informativeness; accurate and complete main concepts produced over the time of discourse elicitation (ACs/min); larger numbers indicate greater efficiency
Picture Naming of untrained items - Boston Naming Test | 3 months
  Change in naming of pictures of untrained items; 60 pictured items; higher score indicates improvement
Naming Response Time of untrained items - Boston Naming Test | 3 months
  Change in response time of naming of pictures of untrained items; 0-20 seconds, decreased response time indicates improvement
Naming Efficiency of untrained items - Boston Naming Test | 3 months
  Change in efficiency of naming of pictures of untrained items; median response time divided by proportion correct naming; smaller numbers indicate greater efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Richardson, Ph.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Center for Brain Recovery and Repair, Albuquerque, New Mexico, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04432883/ICF_000.pdf